CLINICAL TRIAL: NCT00209365
Title: The Role of Pollen Starch Granules in Pollen Challenge Studies in the Fraunhofer Environmental Exposure Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 04/07 Starch granules ITEM
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Asthma; Seasonal Allergic Rhinitis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic, Seasonal

INTERVENTIONS:
Procedure: exposure to grass pollen/starch granules

SUMMARY:
The aim of the study is to explore the contribution of pollen starch granules to the induced symptoms and airway inflammation in patients with allergic rhinitis and mild asthma in a controlled pollen exposure(pollen challenge room at the Fraunhofer ITEM). Starch granules are released from the pollen grains and are considered to be the allergen carriers of the pollen. The hypothesis is proposed that pollen starch granules are important in the induction of airway inflammation and airway hyperresponsiveness.

ELIGIBILITY:
Inclusion Criteria:

* • Male and female subjects, aged 18-55 years. Women will be considered for inclusion if they are:

  * Not pregnant or nursing.
  * Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal with documented proof of hysterectomy or tubal ligation, or meet clinical criteria for menopause and have been amenorrhoeic for more than 1 year prior to the screening visit).
  * Of childbearing potential and using an appropriate method of contraception (Oral contraceptive pill or double barrier).
  * Documented history of bronchial asthma first diagnosed at least 6 months prior to the screening visit and currently being treated only with intermittent short-acting beta2-agonist therapy by inhalation. Patients on low dose steroids will be washed out for 4 weeks.
  * FEV1 > 80% of predicted at screening.
  * They have history of allergic rhinitis to grass pollen and a positive skin prick test for Dactylus glomerata pollen at or within 12 months prior to the screening visit.
  * Documented sensitivity to AMP with a provocative concentration of AMP resulting in a 20% fall in FEV1 (PC20 AMP) of <80mg/ml at the screening visit.
  * Non smoker or smokers with a history of less than 10 pack years.
  * Able and willing to give written informed consent to take part in the study.
  * Available to complete all study measurements.

Exclusion Criteria:

* • History of a respiratory tract infection and/or exacerbation of asthma within 4 weeks before the informed consent and during the study.

  * Any history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnoea, respiratory arrest or hypoxic seizures.
  * Administration of oral, injectable or dermal corticosteroids within 8 weeks or intranasal and/or inhaled corticosteroids within 4 weeks of the screening visit.
  * Administration of xanthines (including theophylline, but not including caffeine), anticholinergics, cromoglycates and/or long acting beta-agonists within 1 week of the screening visit.
  * Unable to abstain from other medications including non-steroidal anti-inflammatory drugs (NSAIDS), anti-depressant drugs, anti-histamines and anti-asthma, anti-rhinitis or hay fever medication (other than short acting inhaled beta-agonists) and paracetamol (up to 1g paracetamol per day is permitted for the treatment of minor ailments e.g. headache) for 1 week prior to screening and throughout the course of the study.
  * Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis). History of MI or CVA are specific contra-indications to AHR testing
  * Known or suspected hypersensitivity or adverse reaction to AMP
  * Subject is undergoing allergen desensitisation therapy
  * There is a risk of non-compliance with study procedures
  * Neurological or psychiatric disease or history of drug or alcohol abuse which would interfere with the subject's proper completion of the protocol assignment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24
Dates: Start 2005-09; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
AMP hyperrespnsiveness

SECONDARY OUTCOMES:
exhaled NO
FEV1
Rhinomanometry

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Krug, MD, Principal Investigator — Fraunhofer ITEM
Locations (1):
- Fraunhofer ITEM, Hanover, Germany